CLINICAL TRIAL: NCT01569321
Title: Diagosis of Breast Carcinoma: Characterization of Breast Lesions With CLEARPEMSONIC : Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011-A01673-38; 2011-40 (Other: AP HM)
Record Dates: First submitted 2012-03-23; First posted 2012-04-03 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast cancer (Experimental)
  Interventions: Device: MRI; Device: PET-CT scan; Device: PEM scan with ClearPemSonic

INTERVENTIONS:
Device: MRI
Device: PET-CT scan
Device: PEM scan with ClearPemSonic

SUMMARY:
Breast cancer is the first cancer in women, the second etiology of death by cancer and the first cause for women between 35 and 55 years.

Diagnostic tools and large screening have been realized with positive impact in a recent review with 31% less likely to die of breast cancer over nearly 30 years compared to women who didn't get regular screening mammograms. Diagnostic tools and treatment also are improving continuously.

However, for some women, breast cancer diagnosis is difficult, in case of high density breast, breast modifications after surgery… In these cases, breast MRI is currently the best imaging tool, with high sensitivity about 90% but with a lower specificity about 60%, that lead to futile biopsies.

Recently, molecular imaging with PET-CT scan with 18FDG has permitted to widely modify cancer treatment.

However, PET-CT scan is not a good imaging tool for initial diagnostic of breast tumor because of a lack in spatial resolution about 8mm. So, researchers developed dedicated PET scan for breast, called Positron Emission Mammography. Our project is in this field of view and is named CLEARPEMSONIC.

First clinical studies with PEM showed very good performance of this imaging modality for initial evaluation of breast tumors. PEM performance is not affected by breast density, hormonal status. Spatial resolution is less than 3mm. PEM seems complementary with MRI, adding a better specificity value.

In the field of CERIMED, ClearPemSonic Project aims to evaluate an new imaging tool which combined PEM scan and ultrasonography.

Technologic evaluation was made. Now a feasibility study is the first step for clinical applications.

The main objective of this project is to confirm the feasibility of PEM scan with the ClearPEmSonic.

Secondary objectives are to compare results with other conventional imaging modalities and MRI.

The gold standard will be histology of the breast tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Mammary Néoplasia ready(in position) (diagnosed on histological taking of type(chap) biopsy)
* Waits whose realization of an imaging TEP-TDM in the 18FDG is required for the coverage(care) of a mammary néoplasia. The decision of realization of this TEP-TDM can be validated during a RCP.

Exclusion Criteria:

* Other cancerous affection;
* Pregnant Woman. Nursing mother
* Patient presenting difficulties of follow-up (insufficient motivation, imminent transfer(transformation) in a city where the study cannot be led)
* Patient incapable to give their written consent.
* Patient claustrophobic or presenting a contraindication to the realization of the MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
MEASURE the Positron Emission Mammography (PEM) | 12 months
  the feasibility of PEM scan with the ClearPEmSonic

SECONDARY OUTCOMES:
MEASURE the other conventional imaging modalities and MRI. | 12 MONTHS
  to compare results with the different device

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France